CLINICAL TRIAL: NCT05497882
Title: Computer-based Learning to Enhance ADRD Care in Prison: Just Care for Dementia
Brief Title: Computer-Based Learning to Enhance Dementia Care in Prison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 336/NOT a clinical trial; R41AG078103 (NIH)
Record Dates: First submitted 2022-07-27; First posted 2022-08-11 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Dementia; Prisoners
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: this is not a clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training Prototype (Experimental): Testing of 3 e-learning modules
  Interventions: Behavioral: E-Learning Prototype for Dementia Care

INTERVENTIONS:
Behavioral: E-Learning Prototype for Dementia Care — Usability testing System Usability Scale

SUMMARY:
The mission of corrections is to provide care, custody, and control for incarcerated individuals. United States prisons are required by law to provide adequate care for growing numbers of older people who are incarcerated-a group who are disproportionately at risk for Alzheimer's Disease and Related Dementias (ADRD). This Phase I project focuses on research and development of highly interactive computer-based learning modules, for prison staff and people who are incarcerated and serving as peer caregivers, to promote an integrated systems approach for enhancing the care of people with ADRD in prison.

DETAILED DESCRIPTION:
U.S. prison systems face sharply increased demands in caring for older people living in prisons. Alzheimer's Disease and related dementias (ADRD) are age-related diseases. Prison populations are over-represented by minority populations who experience disparities in prevalence and incidence of dementia. Prison health, social, and security staff perceive they lack the skills and knowledge essential for identifying dementia and supporting people who are incarcerated and living with ADRDs. This unmet need may be due to a lack of standardized, feasible, and acceptable ADRD education programs that are tailored specifically for those managing and caring for people in the restrictive environment of prisons. Some prisons engage carefully vetted incarcerated people to be peer caregivers, assisting staff with care for people with ADRD. Training programs in prisons are often homegrown and lack consistency, which points to a need for evidence-based, current, and readily accessible training for both prison staff and peer caregivers that is focused on the care of people who are living with ADRD in prison. In response to this need, this Phase I Small Business Technology Transfer project, titled Computer-based Learning to Enhance ADRD Care in Prison: Just Care for Dementia, will demonstrate the scientific merit and feasibility of developing media-rich learning modules to train both multidisciplinary prison staff and peer caregivers on topics related to ADRD care. The specific aims of the project are to (1) transform best practices in ADRD care into media-rich, highly interactive, computer-based educational module prototypes to prepare corrections staff and peer caregivers to meet the growing care needs of people who are incarcerated and living with ADRD; and (2) conduct in-person usability testing of the learning module prototypes with corrections staff and peer caregivers to evaluate the user interface, ease of use, and perceived barriers in order to refine the product and optimize implementation in prison settings. In collaboration with an advisory board comprised of people with expertise in prison healthcare, training and technology, dementia in prisons, and experience with previous incarceration, the investigators will plan and develop discussion guides and then conduct focus groups with two groups of prison stakeholders: interdisciplinary corrections staff and inmates who serve as peer caregivers at a men's and a women's prison. Focus groups will ensure that design and technology plans match what is allowable for training in prison settings and will isolate essential ADRD content for the development of the comprehensive training program. Finally, the investigators will create and evaluate prototypes of media-rich, interactive computer-based learning modules for corrections staff and peer caregivers. At the end of Phase I, the investigators will have: a specifications document for the design of modules that at once fits with the technology available in corrections settings; is permissible to be used by people who are incarcerated; represents the critical learning needs of corrections staff and peer caregivers for providing ADRD care, and further develop collaborative relationships in preparation for commercialization of the product.

ELIGIBILITY:
Inclusion Criteria:

Prison staff:

* work at a participating prison;
* care for or manage people with ADRD in prison;
* able to speak, understand and read English;
* able to consent.

Inmates:

* have experience in caregiving;
* able to speak, understand and read English;
* able to consent.

Exclusion Criteria:

Prison staff:

* not work at a participating prison;
* do not care for or manage people with ADRD in prison;
* cannot speak, understand or read English,
* unable to consent.

Inmates:

* do not have experience in caregiving;
* cannot speak, understand or read English,
* unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Focus Groups | Focus groups will conducted in year 1. The analysis will be completed in Year 1 immediately following the conduct of the focus groups.
  Focus groups will be conducted with interdisciplinary staff and peer caregivers. Data evaluation will include content and thematic analysis using constant comparative analyses methods.
System Usability Scale | The usability test will be conducted in Year 1 and system usability scale will be administered in Year 1 following the conduct of the usability test.
  The System Usability Scale is a validated tool for assessing the usability and acceptability of technological products. Items on the System Usability Scale are rated from 1 (minimum) to 5 (maximum) with the higher number representing the better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Loeb, Principal Investigator — Penn State University
Locations (2):
- United States (2):
  - Barbara Walkosz, Golden, Colorado
  - Penn State University, University Park, Pennsylvania